CLINICAL TRIAL: NCT03861754
Title: Effects of Physical Activity on Weight Loss and Weight Maintenance in Obese Adults - Three Year Follow-up Study
Acronym: LILA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu Deaconess Institute Foundation sr (Unknown); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Kaisu Kaikkonen, Researcher, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147/2006
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Weight Loss; Physical Activity; Healthy Obesity, Metabolically
Keywords: Obesity; Weight loss; Weight maintenance; Physical activity; Fitness
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity; Obesity, Metabolically Benign

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lifestyle modification (Experimental): intensified Behavioural Modification (iBM) group receiving lifestyle counselling
  Interventions: Behavioral: Lifestyle modification
- Lifestyle modification and exercise 1 (Experimental): Intensified Behavioural Modification and exercise from 0 to 3 months (CWT1) group:
  Lifestyle counselling 3 months Exercise intervention from 0 to 3 months
  Interventions: Behavioral: Lifestyle modification
- Lifestyle modification and exercise 2 (Experimental): Intensified Behavioural Modification and exercise from 6 to 9 months (CWT2) group:
  Lifestyle counselling 3 months Exercise intervention from 6 to 9 months
  Interventions: Behavioral: Lifestyle modification
- Control Group (No Intervention): Control group, no intervention, only measurements and questionnaires

INTERVENTIONS:
Behavioral: Lifestyle modification
  Other Names: Lifestyle modification and exercise 1; Lifestyle modification and exercise 2
  Arms: Lifestyle modification; Lifestyle modification and exercise 1; Lifestyle modification and exercise 2

SUMMARY:
Objective To study if exercise added to weight loss treatment at the beginning of the weight loss intervention or at 6 months could sustain the weight loss achieved or give extra boost for weight reduction.

Design 36-month, 4-group parallel, randomized trial.

Setting Oulu, Finland.

Participants 120 obese adults (body mass index ≥ 30).

Intervention Participants were randomly assigned to behavioural modification (iBM) (n = 30), behavioural modification + exercise from 0 to 3 months (CWT1) (n = 30), behavioural modification + exercise from 6 to 9 months (CWT2) (n = 30), and a control group (CON) (n = 30). Questionnaires and measurements were performed at baseline, 3,9,4 and 36 months. The intervention consisted of an intensified weight loss period (1-12 months) followed by a weight maintenance period (13-36 months). Intensified behavioural modification included 14 individual face to face meetings, eleven times with a personal therapist (qualified nurse) and three times with a nutritionist. Weight maintenance period included six individual meetings with personal therapist. Twelve weeks supervised exercise was offered three times a week, 40 minutes at a time. In the CWT1 group supervised exercise was offered at months 1-3 and in the CWT2 group at months 4-6.

Measurements Body weight (primary outcome) and waist circumference (secondary outcome)

ELIGIBILITY:
Inclusion Criteria:

* Body mass Index > 30
* Age 18-64

Exclusion Criteria:

* Pregnancy
* Health reasons preventing exercise and exercise test
* Medication preventing exercise and exercise test
* Previously diagnosed diabetes

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2004-01-28 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Weight change | Change from baseline weight at 36 months
  Kilograms

SECONDARY OUTCOMES:
Waist circumference change | Change from baseline waist circumference at 36 months
  Cm

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu Deaconess Institute Foundation sr, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No